CLINICAL TRIAL: NCT03325413
Title: Improvement of Perioperative Care of Elderly Patients
Acronym: PeriAge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: PV5596; 01VSF16057 (Other Grant/Funding Number: DLR German Aerospace Center)
Record Dates: First submitted 2017-10-02; First posted 2017-10-30 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Perioperative Care
Keywords: Perioperative geriatric care; Geriatric assessment; Postoperative cognitive dysfunction; POCD; Frailty; Depression; Physical fitness; Geriatric anesthesia; IADL; Postoperative functional status; Quality of life
MeSH Terms: conditions — Postoperative Cognitive Complications; Frailty; Depression | interventions — Restraint, Physical; Breathing Exercises; Dietary Supplements; Anesthesia, Conduction; Hypothermia, Induced

STUDY DESIGN:
Intervention Model Description: The study has 3 arms with patients allocated to them in a fixed chronological order.
  For six months, patients will be recruited for the control arm. In this arm, participants receive usual care without any additional intervention initiated by the study.
  After finishing recruitment for the control arm, patients will be recruited for the implementation arm for six months. In this arm, stepwise implementation of the study interventions begins with the possibility of flexibly adapting them to the specific conditions.
  After finishing recruitment for the implementation arm, patients will be recruited for the full-scale intervention arm for six months. In this arm, all study interventions will be utilized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Usual care with assessment only (no study-related intervention)
- Implementation (Other): Implementation of intervention measures
  Interventions: Behavioral: Systematic inclusion of family members; Behavioral: Preoperative information; Behavioral: Physical and breathing exercises; Dietary Supplement: Dietary supplements; Other: Evaluation of long-term medication; Procedure: Regional anesthesia; Other: Personal aids; Device: Temperature management; Device: Neurmonitoring; Procedure: Pain catheter
- Full-scale intervention (Other)
  Interventions: Behavioral: Systematic inclusion of family members; Behavioral: Preoperative information; Behavioral: Physical and breathing exercises; Dietary Supplement: Dietary supplements; Other: Evaluation of long-term medication; Procedure: Regional anesthesia; Other: Personal aids; Device: Temperature management; Device: Neurmonitoring; Procedure: Pain catheter

INTERVENTIONS:
Behavioral: Systematic inclusion of family members — Systematic inclusion of family members/ reference person in the perioperative process
  Arms: Full-scale intervention; Implementation
Behavioral: Preoperative information — Detailed preoperative information about delirium prevention and procedures
  Arms: Full-scale intervention; Implementation
Behavioral: Physical and breathing exercises — Preoperative execution of physical and breathing exercises if necessary
  Arms: Full-scale intervention; Implementation
Dietary Supplement: Dietary supplements — Dietary supplements if necessary
  Arms: Full-scale intervention; Implementation
Other: Evaluation of long-term medication — Avoidance of unsuitable drugs for elderly if possible
  Arms: Full-scale intervention; Implementation
Procedure: Regional anesthesia — Regional anesthesia whenever possible
  Arms: Full-scale intervention; Implementation
Other: Personal aids — Personal orientation aids until anesthesia induction
  Arms: Full-scale intervention; Implementation
Device: Temperature management — Perioperative warming
  Arms: Full-scale intervention; Implementation
Device: Neurmonitoring — Using Bispectral index (BIS) to measure the depth of anesthesia
  Arms: Full-scale intervention; Implementation
Procedure: Pain catheter — A pain catheter will be used as postoperative pain therapy if possible
  Arms: Full-scale intervention; Implementation

SUMMARY:
The focus of this study is the development of a perioperative treatment concept for elderly patients, based on individual necessities and risk factors, aiming to improve patient outcome. The planned interventions include preoperative screening for malnutrition, frailty and uncalled-for long-term medication, if required followed by early prophylaxis and treatment of these risk factors, prior to or during surgery.

DETAILED DESCRIPTION:
In Germany every second inpatient surgical intervention is performed on patients aged 60 years and above. These patients often offer an extensive set of risk factors such as frailty, malnutrition, poor physical fitness and multi-morbidity that may in turn lead to longer hospitalizations and decline of health and functional status after surgery. An age-related increase in postoperative complications, such as postoperative cognitive dysfunction (POCD) and delirium is associated with a higher rate of postoperative morbidity, mortality and longer hospitalization.

Early detection of risk factors and implementation of prophylactic measures is important to reduce postoperative complications and improve clinical outcomes in elderly patients. The aim of our study is to develop and verify a protocol - which allows for a systematic evaluation of risk factors and the implementation of prophylactic or therapeutic measures in order to optimize the postoperative outcome. The feasibility of our protocol will be verified in clinical practice by systematic process evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Age >64 years
* Written informed patients consent
* forthcoming elective surgery
* Time interval from inclusion to appointed surgery at least 5 days

Exclusion Criteria:

* Refusal of consent
* Illiteracy
* Poor knowledge ofGerman language
* Mental disability
* Vision handicap (not corrected)
* Hearing handicap (not corrected)
* Benzodiazepine abuse
* Drug/ substance abuse
* Psychosis
* Parkinson disease
* Emergency surgery
* Planned postoperative ICU treatment
* Planned inpatient stay 1 night
* Cerebral surgery
* Ophthalmological surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 310 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-05-14 (Actual); Study Completion 2020-05-14 (Actual)

PRIMARY OUTCOMES:
Functional abilities | Evaluation preoperatively, 1 month, 6 months after surgery
  Change in functional abilities from baseline, evaluated by Instrumental Activities of Daily Living (IADL) score

SECONDARY OUTCOMES:
Cognitive impairment | Evaluation preoperatively, at 2-5 days, 1 month, 6 months after surgery
  DemTect: cognitive screening instrument, sensitive to the early symptoms of dementia
Attention and task switching | Evaluation preoperatively, at 2-5 days, 1 month, 6 months after surgery
  The Trail Making Test A&B (TMT A&B): a neuropsychological test of visual attention and task alternation
Attentional capabilities | Evaluation preoperatively, at 2-5 days, 1 month, 6 months after surgery
  TAP Alertness: a computerized, standardized neuropsychological test for attentional performance.
Health related quality of life | Evaluation preoperatively, 1 month, 6 months after surgery
  Measured by a 12-item short-form (SF-12) Health Survey
Hospital length of stay | 1 month
  Day of admission until day of discharge
Postoperative complications | Evaluation evaluation of complications at 2-5 days, 1 month, 6 months after surgery
  Incidence of postoperative complications

OTHER OUTCOMES:
Quality of delivery of the intervention components | 6 months
  Continuous documentation of which intervention components were delivered by the clincal staff with a standardized checklist
Experience of staff with intervention components | 6 months
  Qualitative interviews with the clinical staff on acceptability, feasibility, barriers, and facilitators of the intervention
Mobility | Evaluation preoperatively, 1 month, 6 months after surgery
  Timed Up&Go-Test
Physical fitness | Evaluation preoperatively, 1 month, 6 months after surgery
  Sit-to-stand- Test
Grip strength | Evaluation preoperatively, at 2-5 days, 1 month, 6 months after surgery
  Measurement by Vigorimeter
Frailty | Evaluation preoperatively and 6 months after surgery
  LUCAS (Longitudinale Urbane Cohorten Alters - Studie) functional Index
Mental Health | Evaluation preoperatively, 1 month, 6 months after surgery
  Geriatric Depression Scale (GDS) by Yesavage: a 15-item self-report assessment used to detect depression in the elderly

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology and Intensive Care Medicine, University Medical Center Hamburg-Eppendorf (UKE), Hamburg, Germany

REFERENCES:
- [Derived] Lebherz L, Olotu C, Koch B, Kiefmann R, Harter M, Kriston L. Evaluating the implementation process of a multicomponent perioperative intervention for prevention of postoperative functional decline in geriatric patients: a qualitative study. BMJ Open. 2025 Dec 18;15(12):e104460. doi: 10.1136/bmjopen-2025-104460. PMID 41412625
- [Derived] Olotu C, Lebherz L, Mende A, Hempel C, Philipp R, Schroeter J, Plumer L, Koch B, Harter M, Zollner C, Kriston L, Kiefmann R. Feasibility and effectiveness of an evidence-based intervention bundle to improve peri-operative care of older adults: A quality improvement study. Eur J Anaesthesiol Intensive Care. 2024 Jul 4;3(4):e0055. doi: 10.1097/EA9.0000000000000055. eCollection 2024 Aug. PMID 39917250
- [Derived] Olotu C, Lebherz L, Harter M, Mende A, Plumer L, Goetz AE, Zollner C, Kriston L, Kiefmann R. Improvement of perioperative care of the elderly patient (PeriAge): protocol of a controlled interventional feasibility study. BMJ Open. 2019 Nov 24;9(11):e031837. doi: 10.1136/bmjopen-2019-031837. PMID 31767591